CLINICAL TRIAL: NCT07265583
Title: Electrical Impedance Tomography and Lung Ultrasound Score in Early Prediction of Bronchopulmonary Dysplasia in Preterm and Very Low Birth Weight Infants.
Brief Title: Early Prediction of Lung Injury in Preterm Infants Score
Acronym: EPLIPS
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Ghirardello, MD, Chief of Neonatal Unit and Neonatal Intensive care Unit, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: EPLIPS
Record Dates: First submitted 2025-09-09; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Distress Syndrome RDS; Preterm Birth
Keywords: Respiratory distress syndrome RDS; preterm neonate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The main hypothesis is that even preterm infants considered "stable" receiving non-invasive ventilation may be at risk of developing BPD due to an inhomogeneous distribution of ventilation. Identifying this characteristic from the first days of life by using EIT could, in the future, optimize non-invasive ventilation strategies as early as possible, such as lung recruitment manoeuvres, which are currently mainly used during invasive mechanical ventilation. In addition, comparing the LUS scores and homogeneity parameters derived from the EIT may help to further confirm the role of semi-quantitative lung ultrasound as a rapid, non-invasive, and readily available tool in NICUs for monitoring the lung function of preterm infants in the short and long term.

The primary objective is to measure homogeneity by Electrical Impedance Tomography (EIT) technology, used in the first weeks of life, for the development of BPD of grade 3, at 36 weeks postmenstrual age or death, in stable preterm infants requiring non-invasive ventilation. The secondary objective are to score if homogeneity at EIT are present and whether if they are associated with BPD. to ompare the distribution of regional lung ventilation obtained by EIT with the validated LUS scores.

DETAILED DESCRIPTION:
104 preterm infants born between 26 and 32 weeks of gestational age and/or with a birth weight < 1500g (very low birth weight infants - VLBW) with respiratory distress syndrome (RDS). are enrolled in the study In non-invasive ventilation (nasal continuous positive airway pressure -nCPAP- or high flow nasal -HFNC-) at 72h of life.

The study will be conducted at the Neonatal Intensive Care Unit of the Fondazione Policlinico San Matteo IRCSS,Pavia, Italy; PI Dr. S. Ghirardello; Chief of NICU.. Participation at the study will not modify the standard clinical care. In particular, the data obtained from this study will not be used to change the clinical practice in use at the time of the study and the investigators will supervise the proper conduct of the research.Recruitment of patients will be consecutive and continuous through the project investigator in daily clinical practice, if the criteria for inclusion in the study will be met and after obtaining informed consent from the parents.

The study procedures follow the standard clinical practice at our Unit, inclusive of lung ultrasound (LUS). In addition, Electrical Impedance Tomography (EIT) will be performed.

Briefly, after stabilization in delivery room, the clinicians start nCPAP or HFNC and administer surfactant therapy, according to "European guidelines 2022" and standardized internal protocols. The surfactant therapy should be given early in the course of the disease. The suggested protocol would be to treat worsening babies with RDS when FiO2 > 0.30 on CPAP pressure ≥6 cm H2O or if lung ultrasound suggests surfactant need. Less invasive surfactant administration (LISA) is the current preferred method of surfactant administration for spontaneously breathing babies on CPAP. The decision to intubate and start endotracheal mechanical ventilation (MV) is based on the development of respiratory acidosis (pH < 7.20, pCO2 > 60-65mmHg) or severe apnea. While on MV, the SatO2 target was 90%-94%; pH is kept between 7.25 and 7.35, and pCO2 is maintained between 45 and 60mmHg as per local protocols. Infants will be extubated if mean airway pressure (MAP) < 8 cmH20, FiO2 < 0.30, and good respiratory drive is evident.

EIT ENLIGHT 2100 (Timpel®) is a bedside system that uses high-frequency, low-intensity electric signals to provide live images of the breathing lung showing pulmonary performance in real-time. The specific neonatal 16-electrode bands made of hypoallergenic material, soft and thin, will be applied to the chest at the nipple level and will be connected to the tomograph for 60 minutes. During each intervention period, four 10-minute EIT sequences are recorded and for each recording, the first 30 stable consecutive breaths of artefact-free tidal ventilation will be identified. EIT recordings will be made after allowing the infant to stabilize, and in supine position. The raw EIT data will be reconstructed according to standardized guidelines with an anatomically correct and customized human chest algorithm using the manufacturer's software package to exclude impedance variations outside the boundaries of the left and right lungs. Once reconstructed, each of the recordings will be manually examined. Functional EIT images of the current volume distribution will be created, and data extracted from the entire lung, the right and left lungs.

The net signal at end-expiration (end-expiratory lung impedance; EELI) is isolated as the impedance signal at the end of each expiration in arbitrary units to assess overall lung aeration. This is determined in the whole lung (EELI total) and in four regions of interest (ROIs): horizontal quantiles ranging from non-gravity dependent (NGD) to gravity dependent (GD) lung fields (EELINGD, EELImidNGD, EELImidGD, EELIGD) to assess global and regional aeration. Homogeneity of lung aeration during non-invasive ventilation will be measured. To do this, signals in each quantile of regional aeration will be first weighted to the known pixel contribution of each region to normalise for differences in lung size. Then, the NGD half of the EIT signal will be divided by the GD half:

Aeration homogeneity ratio (AHR) = EELINGD +EELI mid NGD/ EELIGD +EELI mid GD A value of 1 represents equal distribution of air and a value <1 or >1 describes an aeration which favours the GD or NGD lung, respectively.

As per study protocol, electrical impedance tomography will be applied following specific timing: the first one (T0) is performed at 72 h of life, the second one (T1) at seven days of life, and the last one at 14 days of life (T2).

At the same time points, lung ultrasound will be performed. Images are obtained with a Hitachi Arietta v70 ultrasound scanner. A linear probe (5-12 MHz) is used. Trained physicians perform the LUS and assign the nLUS score. According to the study by Brat et al., each lung is divided into three areas, and a score from 0 to 3 was given to each scan. 0 indicates A-pattern (defined by the presence of only A-lines); 1 indicates B-pattern (i.e., alveolar-interstitial pattern, described as the presence of at least three well-spaced B lines); 2 indicates severe B-pattern (i.e., severe alveolar-interstitial pattern, defined as the presence of crowded and coalescent B-lines with or without subpleural consolidations with a depth < 1 cm); and 3 indicates consolidation (i.e., subpleural echo-poor or tissue-like echotexture area with depth > 1 cm and irregular borders, which may also have mixed hypoechogenic and hyperechogenic spots representing air bronchograms). Therefore, a total score from 0 to 18 is assigned to the LUS.

The exams will be performed after the patient's standard care to minimize neonatal discomfort. Peripheral capillary oxygen saturation (SpO2) and heart and respiratory rate (RR) are measured continuously.

ELIGIBILITY:
Inclusion Criteria: preterm infants born between 26 and 32 weeks of gestational age and/or with a birth weight < 1500g (very low birth weight infants - VLBW) with respiratory distress syndrome (RDS).

- Exclusion Criteria: - outborn infants

* complex congenital malformations
* metabolic, chromosomal, or other genetic abnormalities
* pulmonary hypoplasia, congenital anomalies of surfactant proteins or other pulmonary abnormalities
* any skin anomalies
* need for mechanical ventilation > 72h after birth
* any life-threatening comorbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.
* lack of parent consent.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For this study we will enrol 104 preterm infants born between 26 and 32 weeks of gestational age and/or with a birth weight < 1500g (very low birth weight infants - VLBW) with respiratory distress syndrome (RDS). The patients are considered eligible to be enrolled in the study if they are assisted in non-invasive ventilation (nasal continuous positive airway pressure -nCPAP- or high flow nasal -HFNC-) at 72h of life.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The prognostic value of homogeneity of ventilation assessed with EIT | 24 months
  The primary objective is to measure the benefit of an earlier detection of the risk to develop BPD at 36 weeks postmenstrual age in stable preterm infants requiring non-invasive, in the first weeks of life, scoring the homogeneity of ventilation using EIT technology ventilatio measured by EIT technology, used in the first weeks of life, for the development of BPD at 36 weeks postmenstrual age

SECONDARY OUTCOMES:
changes in homogeneity at EIT | 24 months
  to measure whether changes in homogeneity at EIT are present (YES/NO)
homogeneity at EIT are associated with BPD or death | 24 months
  Score changes in homogeneity at EIT and association to BPD or death
EIT and LUS score | 24 months
  measure the association of the distribution of regional lung ventilation obtained by EIT with the validated LUS scores

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ghirardello, MD, Principal Investigator — NICU, Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy